CLINICAL TRIAL: NCT04564287
Title: An Observational Study of Neurologic Function After COVID -19 Infection
Brief Title: An Observational Study of Neurologic Function After COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000094; 000094-N
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
Keywords: Neurological; COVID-19; Coronavirus; Autonomic; Brain; Natural History
MeSH Terms: conditions — COVID-19; Neurologic Manifestations; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fully Recovered Individuals: Individuals with history of Covid-19 infection who have fully recovered without residual neurological symptoms
- Patients with neuro-PASC: Patients with history of Covid-19 infection and persistent neurological symptoms (Post-Acute Sequelae of SARS CoV-2 Infection, neuro-PASC)

SUMMARY:
Background:

COVID-19 is an infection caused by a coronavirus. It can affect different parts of the body. For most people, it causes fevers or trouble breathing. Some people can have symptoms long after they recover. Researchers want to learn if there are signs of changes in the nervous system that may be related to COVID-19.

Objective:

To test the nervous system (the brain and nerves) in people who have had COVID-19 yet still have certain symptoms even after recovering.

Eligibility:

People age 18 and older who had COVID-19 and still have neurologic symptoms after they recovered from the initial infection.

Design:

Participants will be screened with a medical record review.

Participants will have a neurological exam. They will complete pen-and-paper tests of their memory and thinking. They will complete a smell test with 'scratch-and-sniff' booklets.

They will give blood samples.

Participants will have magnetic resonance imaging (MRI) of the brain. Soft padding or a coil will be placed around their head. They will lie on a table that slides in and out of the MRI scanner. They will get a contrast dye through an intravenous (IV) catheter.

Participants blood pressure, blood flow, skin temperature, sweating, and breathing will be monitored.

Participants will have an electrocardiogram to measure heart function.

Participants will blow into a mouthpiece for several seconds.

Participants will lie on a table that has a motor. The motor tilts the table. Participants will have blood drawn through an IV as the table tilts.

Participants will have a lumbar puncture. A small needle will be inserted into the spinal canal to obtain fluid.

Participants may repeat some tests 8 weeks to 1 year later.

DETAILED DESCRIPTION:
Study Description:

This study will characterize ongoing neurologic abnormalities in those who recovered from acute COVID-19 infection yet have persistent neurologic symptoms. Despite clinical recovery from the acute infection, some individuals continue to experience ongoing symptoms, at times several months after recovery (Post-Acute Sequelae of SARS CoV-2 Infection, PASC), and many of these symptoms are neurologic (neuro-PASC). The NIH Clinical Center provides the breadth of expertise and resources to best investigate this patient group. This study will collect a broad array of specialized neurologic testing in this group who, despite recovering from the acute SARS-CoV-2 infection, continue to experience neurological symptoms. It is hypothesized that this group will have abnormalities on neurologic testing that may identify discrete phenotypes of COVID-19 sequelae. Additionally, by including a group of individuals who have fully recovered without residual neurological symptoms, this study should be able to determine if there are abnormal results of study procedures in the absence of symptoms.

Pre-screening for this study will be done under the study, Post-Coronavirus Disease 19 Syndrome at the National Institutes of Health. Potentially eligible participants will be identified under the screening arm of that study and will be referred to the study team. If deemed eligible for this study based on a review of available records and a telephone discussion with the potential participant, participants may enroll. Enrollment will include a visit to the NIH Clinical Center for informed consent and completion of the study procedures. We anticipate that the baseline study procedures will take approximately 2-3 outpatient visits to complete or the participant may be admitted as an inpatient. Participants may return for an optional follow-up visit (with a repeat of the study procedures done initially) after at least 6 months from completion of their baseline study visit testing.

Objectives:

Primary Objective: To investigate structural brain MRI in those with prior SARS-CoV-2 infection and persistent neurologic symptoms and in those with prior SARS-CoV-2 infection without persistent neurologic symptoms.

Secondary objective:To investigate other components of neurologic function in those with prior SARS-CoV-2 infection and persistent neurologic symptoms and in those with prior SARS-CoV-2 infection and without persistent neurologic symptoms.

Endpoints:

Primary endpoint: The number and character of brain MRI abnormalities on a dedicated research MRI protocol optimized to detect COVID-19-associated disease.

Secondary endpoints:

1. Neurologic examination: The number and character of abnormalities associated with both central and peripheral nervous system disease.
2. Autonomic testing: The number and character of test results indicating autonomic nervous system or catecholaminergic dysfunctions as evidenced by abnormal physiological or neurochemical measures at rest or in response to the Valsalva maneuver or head-up tilting.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in the PASC cohort, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged at least 18 years at the time of enrollment
3. Enrolled in the screening phase of Protocol 000089 Post-Coronavirus Disease 19 Convalescence at the National Institutes of Health
4. Positive COVID-19 test result (per the methodology used for inclusion in Protocol 000089) at least six weeks prior to enrollment and exhibiting persistent neurologic symptoms evidenced by a positive response to at least one of the following:

   1. Do you have ongoing issues with being lightheaded or dizzy and if so, are these issues made worse when you sit or stand up

      quickly?
   2. Do you have ongoing issues with gait instability, problems with vision, speech, swallowing?
   3. Do you have ongoing issues with sensation or strength in your face/arms/legs?
5. Ability of subject to understand and the willingness to sign a written informed consent document.

In order to be eligible to participate in the Fully Recovered cohort, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged at least 18 years at the time of enrollment
3. Enrolled in the screening phase of Protocol 000089 Post-Coronavirus Disease 19 Convalescence at the National Institutes of Health
4. Positive COVID-19 test result (per the methodology used for inclusion in Protocol 000089) in at least six weeks prior to enrollment.
5. A self-reported illness narrative of recovery to prior health after a SARS/CoV2 infection, without residual fatigue, brain fog, orthostatic intolerance, or exercise intolerance.
6. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Presence of a contraindication to research MRI with gadolinium, including contraindicated metal in the body, prior allergic reaction to gadolinium, eGFR <45 mmol/L, pregnancy or lactation, or claustrophobia that is unable to be adequately treated with a low oral dose of a benzodiazepine.
2. Contraindication to a research lumbar puncture, including use of anticoagulant medication, platelets < 50,000/microL, PT or PTT >1.5 x ULN for the NIH Clinical Center, or otherwise inability to complete the procedure.
3. Contraindication to autonomic testing, including refractory ventricular arrhythmias or symptomatic coronary artery disease.
4. A condition prior to the diagnosis of COVID-19 infection that would significantly confound interpretation of the research tests (e.g., prior diagnosis of postural orthostatic tachycardia syndrome), as determined by the study investigators.
5. Fever or respiratory symptoms in the last seven days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
MRI brain | NIH Clinical Center Visit
  The number and character of brain MRI abnormalities on a dedicated research MRI protocol optimized to detect Covid-19-associated disease.

SECONDARY OUTCOMES:
Neurological Examination | NIH Clinical Center Visit
  Neurologic examination: The number and character of abnormalities associated with both central and peripheral nervous system disease.
Autonomic Testing | NIH Clinical Center Visit
  Autonomic testing: The number and character of test results indicating autonomic nervous system disease as evidenced by abnormal heart rate and blood pressure responses during tilt table testing.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000094-N.html